CLINICAL TRIAL: NCT03817268
Title: Capecitabine or Observation for Patients With pT1N+M0 or pT2-3N0M0 Gastric Adenocarcinoma Undergoing R0 Resection (CAPOGA): A Large Multicenter Phase III Randomized Controlled Trial
Brief Title: Capecitabine or Observation for Patients With pT1N+M0 or pT2-3N0M0 Gastric Adenocarcinoma Undergoing R0 Resection
Acronym: CAPOGA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, A-Man Xu, Professor, Chief Surgeon, Department Head, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPOGA-01
Record Dates: First submitted 2019-01-18; First posted 2019-01-25 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capecitabine monotherapy group (Experimental)
  Interventions: Drug: Capecitabine monotherapy
- Control group (No Intervention)

INTERVENTIONS:
Drug: Capecitabine monotherapy — Capecitabine is administered within 6 weeks after resection and after adequate recovery. To reduce the side effects and improve patient compliance, the administered dose is half of the recommendation: 625 mg/m2, bis in die (BID) (1250 mg/m2 per day). A 2-week therapy is followed by a 1-week pause, and a cycle includes 3 weeks. A total of 8 cycles is planned for each patient.
  Arms: Capecitabine monotherapy group

SUMMARY:
Gastric cancer (GC) is one of the most common and lethal malignancies in Asia. For early (stage T1) GC, it has been found by analyzing surgical specimens that ~5% of cancers have lymph node metastasis. For patients with stage T2-3N0M0 GCs, there is a considerable probability of micro-metastasis. While the US National Comprehensive Cancer Network (NCCN), the Japanese Gastric Cancer Association (JGCA), and the European Society for Medical Oncology (ESMO) guidelines recommend adjuvant therapy for most patients with resected >T1N0 GCs, the recommendations vary regarding postsurgical treatment for patients with stage T1N+M0 or T2-3N0M0 disease. The JGCA guidelines do not recommend postsurgical chemotherapy for this patient population, while the ESMO support the adjuvant treatment. The NCCN has not offered a definitive recommendation on this issue. Through careful literature search, there is not yet randomized report on whether postsurgical chemotherapy benefits survival for patients with resected T1N+M0 or T2-3N0M0 GC. The first-line chemotherapy regimen for GC is fluorouracil plus platinum. Among fluorouracil, platinum is especially favored due to its less frequent and less severe adverse effects. This large multicenter phase III randomized controlled trial is led by Department of Gastrointestinal Surgery, The First Affiliated Hospital of Anhui Medical University, and carried out in multiple Chinese centers, aiming to compare the safety and efficacy of capecitabine monotherapy versus no therapy in the adjuvant setting for patients with stage T1N+M0 or T2-3N0M0 GC undergoing R0 Resection.

ELIGIBILITY:
Inclusion Criteria:

* Microscopically-confirmed gastric adenocarcinoma (cardia cancer/adenocarcinoma of the esophagogastric junction);
* Cancer stage pT1N+M0 or pT2-3N0M0;
* Radical R0 resection;
* Retrieved lymph node number ≥15;
* Without hepatic, peritoneal, or other distant metastasis;
* Aged 18-70 years;
* No other cancer-directed therapy except primary cancer resection;
* Good tissue and organ function: white blood cell count ≥4000/mm3; neutrophil count ≥1500/mm3; platelet count ≥100000/mm3; total bilirubin ≤25.7 μmol/L or within 1.5 times the upper threshold; aspartate transaminase (AST) and alanine transaminase (ALT) within 2.5 times the upper threshold; creatinine within 1.25 times the upper threshold; creatinine clearance rate >60 mL/min;
* No serious cardiovascular or cerebrovascular disease;
* No concomitant or previous malignancies;
* Enrolled within 6 weeks after resection;
* Eastern Cooperative Oncology Group (ECOG) score ≤2;
* Clavien-Dindo morbidity score 0-2;
* Patient informed consent.

Exclusion Criteria:

* The need to take phenytoin or coumarin anti-coagulates;
* Allergic to capecitabine or fluorouracil;
* Known DPD activity deficiency (DPYD gene mutation);
* Pregnant or breeding women;
* All others contradictory to the items listed in the Inclusion Criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free/Relapse-free survival | 5 years
  The time interval from randomization to local recurrence/distant metastasis, death, or end of follow-up whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 5 years
  The time interval from randomization to death from any cause or end of follow-up whichever occurs first.
Incidence of Treatment-Emergent Adverse Events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events | 2 years
  Incidence of Treatment-Emergent/Drug-Associated Adverse Events as assessed by National Cancer Institute-Common Terminology Criteria for Adverse Events
Health-related quality of life as assessed by European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-Core 30 | 5 years
  Health-related quality of life as assessed by European Organisation for Research and Treatment of Cancer-Quality of Life Questionnaire-Core 30. Except for the last 2 questions, for the first 28 questions higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided